CLINICAL TRIAL: NCT02065778
Title: A Clinical Study of Autologous Bone Marrow Mononuclear Cells Intrathecal Transplantation in Chronic Stroke
Brief Title: Safety and Efficacy of Autologous Stem Cell Therapy in Chronic Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-08
Record Dates: First submitted 2014-02-15; First posted 2014-02-19 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Biological: Autologous bone marrow mononuclear cell transplantation — bone marrow derived mononuclear cells are administered intrathecally in chronic stroke patients

SUMMARY:
The purpose of this study was to study the safety and effect of stem cell therapy on the functional recovery in patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* above 18 years of age
* diagnosed as stroke by clinical and MRI findings

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever
* hemoglobin less than 8
* bleeding tendency
* bone marrow disorder
* left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, M.S., M.Ch, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Borlongan CV. Bone marrow stem cell mobilization in stroke: a 'bonehead' may be good after all! Leukemia. 2011 Nov;25(11):1674-86. doi: 10.1038/leu.2011.167. Epub 2011 Jul 5. PMID 21727900
- [Derived] Sharma A, Sane H, Gokulchandran N, Khopkar D, Paranjape A, Sundaram J, Gandhi S, Badhe P. Autologous bone marrow mononuclear cells intrathecal transplantation in chronic stroke. Stroke Res Treat. 2014;2014:234095. doi: 10.1155/2014/234095. Epub 2014 Jul 8. PMID 25126443